CLINICAL TRIAL: NCT00772369
Title: Retrospective Safety Survey of Selected Events in the 6 Months Following the 4th Dose of the Pentacel® Vaccination Series in Children
Brief Title: Retrospective Survey of Safety of Fourth Dose Pentacel® in Children
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: M5A08
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Diphtheria; Pertussis; Haemophilus Infection; Tetanus; Polio
Keywords: Pertussis; Whooping cough; Diphtheria; Tetanus; Haemophilus influenzae; Poliovirus Types 1, 2, and 3.
MeSH Terms: conditions — Diphtheria; Whooping Cough; Haemophilus Infections; Tetanus; Poliomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this survey is to collect selected safety data.

Primary Objective:

To collect selected safety data at 6 months following the 4th dose of the Pentacel® series.

DETAILED DESCRIPTION:
This is a retrospective survey to collect selected safety data at 6 months following the 4th dose of Pentacel® in children residing in the Canadian Province of British Columbia who have received the 4th dose of the Pentacel® series before their 2nd birthday.

ELIGIBILITY:
Inclusion Criteria:

* Children residing in the Canadian Province of British Columbia who have received the 4th dose of the Pentacel® series before their 2nd birthday.
* Written Informed Consent and Telephone consent from the parent(s) or guardian(s).
* Able to comply with the survey procedures.

Exclusion Criteria:

* Fourth dose of the Pentacel® series received on or after the child's 2nd birthday.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children residing in the Canadian Province of British Columbia who have received the 4th dose of the Pentacel® series before their 2nd birthday
Sampling Method: Non-Probability Sample
Enrollment: 3214 (Actual)
Dates: Start 2003-09; Primary Completion 2004-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Telephone contact for this study was from 20 September 2003 to 30 April 2004.
Pre-assignment Details: A total of 3214 participants that met the inclusion and exclusion criteria were enrolled in this survey. One participant did not return a record release form and twenty-nine (29) others were also excluded from the Primary Analysis Population because their safety data could not be confirmed.
Groups:
- Study Group: Received 4th dose of the Pentacel® series before 2nd birthday
Period: Overall Study
Arm/Group | Study Group
Started | 3214
Completed | 3213
Not Completed | 1
Not completed — Did not return record release form | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 3214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3214
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.5 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1538
  Male | 1676
Region of Enrollment [Number; unit: participants]
  Canada | 3214

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Positive Response to the Solicited Adverse Events Questionnaire Post 4th Dose of the Pentacel® Vaccination Series
Description: Positive response is a 'Yes' to any of the following questions:
  1. Has your child been admitted to a hospital?
  2. Has your child experienced an illness that made you fear for his/her life (life-threatening episode) that required attendance to the Emergency Room or a Physician's office?
  3. Has your child developed a medical condition that required 3 or more office or emergency room visits for that condition?
  4. Has your child been diagnosed by a physician as having:
  Low blood count or low platelet count? Swelling or redness of the joints? Asthma? Diabetes? Autism?
Time Frame: 6 months post 4th dose vaccination
Population: Participants who completed the whole survey. Those who had confirmed data, or had data that did not require confirmation, or had unconfirmed data.
Measure: Number; unit: Particpants
Arm/Group | Study Group
Number analyzed (Participants) | 3213
Particpants
  Participants with no events reported | 3023
  Participants with events reported and confirmed | 161
  Events at 0 to 180 days after Dose 4 | 149
  Events after Day 180 only | 6
  Events prior to Dose 4 only | 6
  Participants with events not confirmed | 29

2. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAE) Post 4th Dose of the Pentacel® Vaccination Series and Relationship to Study Vaccine.
Description: SAE: any untoward medical occurrence with the following outcomes:
  * death,
  * a life-threatening adverse drug experience (as confirmed by the investigators),
  * inpatient hospitalization or prolongation of existing hospitalization,
  * a persistent or significant disability/incapacity, or
  * a congenital anomaly/birth defect. Medical conditions that required 3 or more office or emergency room visits, and diagnosis by a physician of low blood cell count or low platelet count, swelling or redness of the joints, asthma, diabetes, or autism were also solicited. (MedDRA Version 6.0)
Time Frame: 6 Months post 4th dose vaccination
Population: Response to questionnaire that were confirmed by the primary care physician's office were analyzed, Primary Analysis Population. Unconfirmed safety data form 29 participants were excluded from the primary analysis.
Measure: Number; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 3184
Participants
  SAEs Occurring Post-dose 4 (Any) | 80
  SAEs Occurring Post-dose 4 (Related) | 6
  Red cell aplasia (Any) | 1
  Red cell aplasia (Related) | 1
  Vomiting nos (Any) | 3
  Vomiting nos (Related) | 1
  Difficulty in walking (Any) | 1
  Difficulty in walking (Related) | 0
  Pyrexia (Any) | 2
  Pyrexia (Related) | 1
  Hypersensitivity nos (Any) | 1
  Hypersensitivity nos (Related) | 1
  Bronchiolitis (Any) | 3
  Bronchiolitis (Related) | 0
  Bronchitis viral (Any) | 1
  Bronchitis viral (Related) | 0
  Bronchopneumonia nos (Any) | 2
  Bronchopneumonia nos (Related) | 0
  Cellulitis (Any) | 1
  Cellulitis (Related) | 0
  Croup infectious (Any) | 8
  Croup infectious (Related) | 0
  Gastroenteritis nos (Any) | 6
  Gastroenteritis nos (Related) | 0
  Gastroenteritis rotavirus (Any) | 2
  Gastroenteritis rotavirus (Related) | 0
  Gastroenteritis viral nos (Any) | 2
  Gastroenteritis viral nos (Related) | 0
  Herpes zoster (Any) | 1
  Herpes zoster (Related) | 0
  Kawasaki's disease (Any) | 3
  Kawasaki's disease (Related) | 1
  Lobar pneumonia nos (Any) | 2
  Lobar pneumonia nos (Related) | 0
  Localised infection (Any) | 1
  Localised infection (Related) | 0
  Periorbital cellulitis (Any) | 1
  Periorbital cellulitis (Related) | 0
  Pharyngitis (Any) | 1
  Pharyngitis (Related) | 0
  Pneumonia nos (Any) | 7
  Pneumonia nos (Related) | 0
  Pneumonia viral nos (Any) | 1
  Pneumonia viral nos (Related) | 0
  Tonsillitis viral nos (Any) | 1
  Tonsillitis viral nos (Related) | 0
  Upper respiratory tract infection nos (Any) | 1
  Upper respiratory tract infection nos (Related) | 0
  Urinary tract infection nos (Any) | 1
  Urinary tract infection nos (Related) | 0
  Viral infection nos (Any) | 3
  Viral infection nos (Related) | 0
  Femur fracture (Any) | 1
  Femur fracture (Related) | 0
  Hip dislocation (Any) | 1
  Hip dislocation (Related) | 0
  Diabetes mellitus nos (Any) | 1
  Diabetes mellitus nos (Related) | 0
  Acute lymphocytic leukaemia (Any) | 1
  Acute lymphocytic leukaemia (Related) | 0
  Autism (Any) | 1
  Autism (Related) | 0
  Convulsions nos (Any) | 2
  Convulsions nos (Related) | 0
  Febrile convulsion (Any) | 13
  Febrile convulsion (Related) | 1
  Breath holding (Any) | 1
  Breath holding (Related) | 0
  Balanitis nos (Any) | 1
  Balanitis nos (Related) | 0
  Asthma nos (Any) | 8
  Asthma nos (Related) | 0
  Bronchitis nos (Any) | 1
  Bronchitis nos (Related) | 0
  Pneumonia aspiration (Any) | 1
  Pneumonia aspiration (Related) | 1
  Wheezing (Any) | 1
  Wheezing (Related) | 0

ADVERSE EVENTS:
Time Frame: Safety data were solicited through a retrospective survey within 6 months of the post-4th dose of Pentacel™ vaccine.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 93/3213
Other Adverse Events (participants affected / at risk) | 0/3123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=3213)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (7)
General disorders and administration site conditions (General disorders) | 4 (4)
Immune system disorders (Immune system disorders) | 2 (2)
Infections and infestations (Infections and infestations) | 52 (52)
Injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders (Nervous system disorders) | 18 (19)
Psychiatric disorders (Psychiatric disorders) | 2 (3)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Surgical and medical procedures (Surgical and medical procedures) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.